CLINICAL TRIAL: NCT07310095
Title: Efficacy of Guselkumab in Chinese Participants With Crohn's Disease Following Loss of Response to Ustekinumab
Brief Title: A Study to Evaluate the Efficacy of Guselkumab in Chinese Participants With Crohn's Disease (CD)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNTO1959CRD4007; CNTO1959CRD4007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guselkumab Treatment (Experimental): Participants will receive Guselkumab intravenously (IV) every 4 weeks during the induction phase, followed by subcutaneous (SC) administration of Guselkumab every 4 weeks from Week 12 through Week 44 as maintenance therapy.
  Interventions: Drug: Guselkumab (GUS)

INTERVENTIONS:
Drug: Guselkumab (GUS) — Guselkumab will be administered intravenously or by subcutaneous injection.
  Other Names: TREMFYA

SUMMARY:
The purpose of this study is to evaluate how well guselkumab works in participants with Crohn's disease (CD; a long-term condition causing severe inflammation of the intestinal tract) who no longer respond to treatment with ustekinumab.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of Crohn's disease (CD)
* Diagnosed with active CD, as defined by baseline Crohn's Disease Activity Index (CDAI) score greater than or equal to (>=) 220 and either mean daily stool frequency (SF) count >= 4 or mean daily abdominal pain (AP) score >=2
* Participants had received at least two doses of ustekinumab (UST) (induction of 6 milligram [mg]/kilogram [kg] intravenous [IV] followed by 90 mg subcutaneous [SC] at week 8) as the instruction manual
* Initially responded to UST induction therapy and then lose response to UST
* During the screening period, participants are receiving UST treatment as the first line biologic or second line biologic

Exclusion Criteria:

* Have responded well to treatment with UST in a dosing regime that is not in line with to the approved recommended dosing (for example, multiple intravenous induction) experienced optimized treatment with UST(not as instruction manual)
* Participants with CD requiring urgent surgical or endoscopic intervention, or requiring elective surgery within 2 months
* Is currently enrolled in an interventional clinical study
* Complications of CD, such as symptomatic strictures or stenoses, short gut syndrome
* Have a current or be suspected to have an abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission At Week 48 | At Week 48
  Clinical remission is defined as less than (<) 150-point reduction in Crohn's Disease Activity Index (CDAI) score. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. The CDAI score was assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s), and/or opiates, and general well-being. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Response At Weeks 12, 24 and 48 | At Weeks 12, 24 and 48
  Clinical response is defined as greater than or equal to (>=) 100-point reduction from baseline in CDAI score. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. The CDAI score was assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s), and/or opiates, and general well-being. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Percentage of Participants Achieving Clinical Remission At Weeks 12 and 24 | At Weeks 12 and 24
  Clinical remission is defined as < 150-point reduction in CDAI score. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. The CDAI score was assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s), and/or opiates, and general well-being. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Percentage of Participants Achieving Endoscopic Response | At Weeks 24 and 48
  Endoscopic response is defined as >= 50% improvement from baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) score. The SES-CD is based on the evaluation of 4 variables: (ulcers - scored according to size, proportion of the surface covered by ulcers according to extent, proportion of affected surface with any other lesions according to extent, stenosis [single or multiple, and whether the colonoscopy could pass through the narrow lumen]), each considered in 5 segments of the bowel (the ileum, ascending colon, transverse colon, descending colon, and rectum). An overall total SES-CD score is derived from the sum of all the component scores and can range from 0 to 60. Higher scores indicating severe disease.
Percentage of Participants Achieving Endoscopic Remission | At Weeks 24 and 48
  Endoscopic remission is defined as SES-CD less than or equal to (<=) 2 in any individual component. The SES-CD is based on the evaluation of 4 variables: (ulcers - scored according to size, proportion of the surface covered by ulcers according to extent, proportion of affected surface with any other lesions according to extent, stenosis [single or multiple, and whether the colonoscopy could pass through the narrow lumen]), each considered in 5 segments of the bowel (the ileum, ascending colon, transverse colon, descending colon, and rectum). An overall total SES-CD score is derived from the sum of all the component scores and can range from 0 to 60. Higher scores indicating severe disease.
Baseline Characteristics of Participants With Endoscopic Remission: Age | Baseline
  Baseline characteristics of participants (age) with endoscopic remission will be reported.
Baseline Characteristics of Participants With Endoscopic Remission: Sex | Baseline
  Baseline characteristics of participants (sex) with endoscopic remission will be reported.
Baseline Characteristics of Participants With Endoscopic Remission: Height | Baseline
  Baseline characteristics of participants (height) with endoscopic remission will be reported.
Baseline Characteristics of Participants With Endoscopic Remission: Weight | Baseline
  Baseline characteristics of participants (weight) with endoscopic remission will be reported.
Baseline Characteristics of Participants With Endoscopic Remission: History of Advanced Treatment, Concomitant Medications | Baseline
  Baseline characteristics of participants (history of advanced treatment, concomitant medications) with endoscopic remission will be reported.
Baseline Characteristics of Participants With Endoscopic Remission: Comorbidities | Baseline
  Baseline characteristics of participants (comorbidities) with endoscopic remission will be reported.
Baseline Characteristics of Participants With Endoscopic Remission: Surgeries and Procedures | Baseline
  Baseline characteristics of participants (surgeries and procedures such as apheresis) with endoscopic remission will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Xi'an Janssen Pharmaceutical Clinical Trial, Study Director — Xi'an Janssen Pharmaceutical

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency